CLINICAL TRIAL: NCT02368444
Title: A Cognitive Behavioral Therapy and Yoga Program for Trauma Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Julie Staples, PhD, Assistant Adjunct Professor, Georgetown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITRP-01
Record Dates: First submitted 2015-02-10; First posted 2015-02-23 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Posttraumatic Stress; Sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Group (Experimental): Cognitive Behavioral Therapy and Yoga
  Interventions: Behavioral: Cognitive Behavioral Therapy and Yoga

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy and Yoga — Group Cognitive Behavioral Therapy Treatment and Yoga Program
  Other Names: T.E.A.M. Cognitive Behavioral Therapy; Kundalini Yoga

SUMMARY:
The purpose of the proposed study is to evaluate the effectiveness of a cognitive behavioral therapy (CBT) and yoga program for improving posttraumatic stress disorder (PTSD) symptoms and sleep quality in people who have experienced a traumatic event and are reporting trauma symptoms.

DETAILED DESCRIPTION:
The purpose of the proposed study is to evaluate the effectiveness of a cognitive behavioral therapy (CBT) and yoga program for improving posttraumatic stress disorder (PTSD) symptoms and sleep quality in people who have experienced a traumatic event and are reporting trauma symptoms. The total length of the program will be 8 weeks. The sessions will be held 3 hours per week with 1.5 hours of group cognitive behavioral therapy and 1.5 hours of yoga. Changes in PTSD symptoms and sleep quality will be measured at baseline, immediately following the program, and at 2 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed posttraumatic stress disorder (PTSD) or subthreshold PTSD symptoms

Exclusion Criteria:

* current uncontrolled psychotic or bipolar disorder, significant cognitive impairment, substance dependence, non-English speaking, or a significant medical condition that would interfere with participation in the yoga portion of the program

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in Posttraumatic Stress Symptoms will be measured using the PTSD Checklist for the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) (PCL-5) | Baseline and 8 weeks and 16 weeks
  Changes in Posttraumatic Stress Symptoms will be measured using the PTSD Checklist for the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) (PCL-5)

SECONDARY OUTCOMES:
Changes in Sleep Quality will be measured using the Pittsburgh Sleep Quality Index (PSQI) | Baseline and 8 weeks and 16 weeks
  Changes in Sleep Quality will be measured using the Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Julie K Staples, Ph.D., Principal Investigator — Georgetown University
Locations (1):
- Yoga Studio, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No